CLINICAL TRIAL: NCT03133182
Title: Association of Polypharmacy With Outcomes After Elective Noncardiac Surgery: a Population-based Cohort Study
Brief Title: Polypharmacy and Outcomes After Elective Noncardiac Surgery
Status: Completed | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: DM5
Record Dates: First submitted 2017-04-18; First posted 2017-04-28 (Actual); Results first posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2024-12

CONDITIONS: Polypharmacy; Surgical Procedure, Operative; Morality; Epidemiology
MeSH Terms: interventions — Polypharmacy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Polypharmacy: People taking >=5 unique prescription drugs in the 3 months prior to surgery
  Interventions: Drug: Polypharmacy
- No polypharmacy: People taking <5 unique prescription drugs in the 3 months prior to surgery

INTERVENTIONS:
Drug: Polypharmacy — Patients who are taking >=5 unique prescription drugs in the 3 months prior to surgery
  Groups: Polypharmacy

SUMMARY:
This study investigates the association of preoperative polypharmacy with outcomes and healthcare resource utilization in a population-based sample of older patients enrolled in a universal pharmacare program

DETAILED DESCRIPTION:
Multilevel multivariable regression analysis will be used to investigate the adjusted association between preoperative polypharmacy and postoperative outcomes and healthcare resource utilization. Sensitivity analyses will be used to evaluate the robustness of the primary analysis.

ELIGIBILITY:
Inclusion Criteria:

* Intermediate to high risk elective non-cardiac surgery
* Age >=66 on day of surgery

Exclusion Criteria:

-

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Population-based sample of people having their first eligible surgery during the study period
Sampling Method: Non-Probability Sample
Enrollment: 266499 (Actual)
Dates: Start 2002-04 (Actual); Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McIsaac DI, Wong CA, Bryson GL, van Walraven C. Association of Polypharmacy with Survival, Complications, and Healthcare Resource Use after Elective Noncardiac Surgery: A Population-based Cohort Study. Anesthesiology. 2018 Jun;128(6):1140-1150. doi: 10.1097/ALN.0000000000002124. PMID 29443701

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Polypharmacy | No Polypharmacy
Started | 146029 | 120470
Completed | 146029 | 120470
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Polypharmacy | No Polypharmacy | Total
Number analyzed (Participants) | 146029 | 120470 | 266499
Age, Continuous [Mean (Standard Deviation); unit: years] | 75 (6) | 73 (6) | 74 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81922 | 59512 | 141434
  Male | 64107 | 60958 | 125065
Income quintile [Median (Inter-Quartile Range); unit: Income group] — Neighborhood socioeconomic status of the participants is presented as income quintile (income quintile is a measure of neighbourhood socioeconomic status that divides the population into five income groups (from lowest income to highest income)). The scale is from 1-5 (income group quintile 1 (lowest), 2, 3, 4, 5 (highest)). The groups are based on where 20% of the population falls within each category and therefore values vary by year.
  Income group | 3 [2 to 4] | 3 [2 to 4] | 3 [2 to 4]

OUTCOME MEASURES:

1. Primary Outcome: Mortality
Description: death from any cause
Time Frame: from day of surgery up to 90 days after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Polypharmacy | No Polypharmacy
Number analyzed (Participants) | 146029 | 120470
Participants | 4356 | 1919

2. Secondary Outcome: Complications
Description: Patient with a complication based on clusters of ICD-10 Type 2 codes collected in the hospital record
Time Frame: From day of surgery to day of hospital discharge, up to 365 days after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Polypharmacy | No Polypharmacy
Number analyzed (Participants) | 146029 | 120470
Participants | 31570 | 19815

3. Secondary Outcome: Length of Stay
Description: Number of days in hospital after surgery
Time Frame: date of surgery to date of hospital discharge, or 365 days after surgery, whichever comes first
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Polypharmacy | No Polypharmacy
Number analyzed (Participants) | 146029 | 120470
Days | 5 [4 to 8] | 5 [3 to 7]

4. Secondary Outcome: Costs of Care
Description: Costs related to medical care paid for by the provincial health insurance system
Time Frame: date of surgery up to 90 days after surgery
Measure: Mean (Standard Deviation); unit: Canadian Dollars
Arm/Group | Polypharmacy | No Polypharmacy
Number analyzed (Participants) | 146029 | 120470
Canadian Dollars | 24064 (16624) | 20251 (24424)

5. Secondary Outcome: Institutional Discharge
Description: A discharge location at the end of the surgical episode of care that is not back to the patient's original residence (specifically respite or long term care)
Time Frame: date of surgery to date of hospital discharge, or 365 days after surgery, whichever comes first
Measure: Count of Participants; unit: Participants
Arm/Group | Polypharmacy | No Polypharmacy
Number analyzed (Participants) | 146029 | 120470
Participants | 34128 | 23098

6. Secondary Outcome: Hospital Readmission
Description: Acute hospital readmission after discharge from index hospitalization
Time Frame: From the date of hospital discharge to 30 days after the date of discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Polypharmacy | No Polypharmacy
Number analyzed (Participants) | 146029 | 120470
Participants | 13202 | 8097

ADVERSE EVENTS:
Time Frame: Within 90 days of surgery
Description: All-Cause Mortality: The occurrence of death due to any cause.
  No other adverse events were monitored or reported.
Arm/Group | Polypharmacy | No Polypharmacy
All-Cause Mortality (participants affected / at risk) | 4356/146029 | 1919/120470
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
We are unable to fully account for unmeasured confounders and indication bias. We were not able to account for granular patient-level data. We used health administrative data that were not initially collected for research purposes; risk of misclassification bias should be considered. Our polypharmacy exposure did not account for the potential differing risk impacts or appropriateness of different drugs. We were unable to account for medication underutilization which could bias results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No